CLINICAL TRIAL: NCT06499129
Title: The Effect of Nursing Interventions Based on Levine Conservation Model on Fatigue, Peripheral Neuropathy and Anxiety Levels in Colorectal Cancer Patients Receiving Chemotherapy: A Randomized Controlled Study
Brief Title: LevineConservationModelandColorectalPatients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Collaborators: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Naciye Esra Koyuncu, Researcher Assistant, KTO Karatay University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Necmettin Erbakan University
Record Dates: First submitted 2024-07-01; First posted 2024-07-12 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Fatigue; Peripheral Neuropathy; Anxiety
Keywords: Colorectal cancer, Levine's Conservation Nursing Model, Nursing intervention
MeSH Terms: conditions — Fatigue; Peripheral Nervous System Diseases; Anxiety Disorders; Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trials
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SensoryBall (Experimental): The training content prepared based on the Levine Conservation Model will be given to patients assigned to the intervention group. Training content information in line with the Levine Conservation Model; The conservation model, which is the application of nursing theoretical knowledge for practice, will focus on the applications to be made for three basic principles for the protection of energy, protection of structural integrity and protection of personal integrity.
  Soft plastic sensory balls for hands and feet will be used in the management of peripheral neuropathy symptom.
  In the sensory exercise for the feet, the patient will be asked to place the foot sensory ball between the floor and the foot and roll it to create a slight pressure on the sole of the foot.
  Progressive Relaxation Exercises Practice Progressive relaxation exercises will be played to colorectal cancer patients who will receive chemotherapy.
  Interventions: Behavioral: Sensory ball, progressive relaxation exercise, training
- Control (No Intervention): The control group patients who will receive chemotherapy treatment for the first time and who meet the inclusion criteria will not receive any intervention other than standard chemotherapy treatment and standard nursing care and will be asked to complete the Personal Information Form (only on the first day), Cancer Fatigue Scale, CIPNAT and Trait Anxiety Inventory on the first chemotherapy day, 14th day and 28th day.

INTERVENTIONS:
Behavioral: Sensory ball, progressive relaxation exercise, training — The effect of sensory ball use on fatigue, peripheral neuropathy and anxiety will be examined
  Arms: SensoryBall

SUMMARY:
Colorectal cancer is one of the most common types of cancer in the world, ranking 3rd among cancers that cause death in men and women. In patients diagnosed with colorectal cancer, chemotherapy treatment is planned to prolong survival as in all other cancer patients. Among the side effects of chemotherapy treatment, it is known that fatigue develops between 50-90%, which is mild for one week in 45% of patients and persists for two weeks in 33%. In the literature, the incidence of chemotherapy-induced peripheral neuropathy is reported to be between 10-100% depending on the type and dose of the drug taken. Alejandro et al. (2013) reported that the incidence of oxaliplatin-related peripheral neuropathy was 84%, which was acute in 74% of patients and permanent in 48%. In addition, anxiety disorders are among the common mental symptoms in cancer patients and their prevalence has been reported to be 10-30%.

In this study, it is aimed to reveal the effect of nursing interventions based on Levine's Conservation Model on fatigue, peripheral neuropathy and anxiety levels in colorectal cancer patients receiving chemotherapy treatment.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-75
* Diagnosed with primary and new colorectal cancer (Stage II and III),
* The decision to start the FOLFOX treatment protocol has been taken,
* Having a smartphone,
* Being literate,
* Ability to speak and understand Turkish,
* Open to communication and cooperation.

Exclusion Criteria:

* History of neuropathy or diabetes,
* History of hypothyroidism, renal failure,
* Hearing, speech and vision problems,
* Receiving radiotherapy or immunotherapy,
* Psychiatric diagnosis or ongoing treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2025-06-25 (Actual); Primary Completion 2025-12-28 (Actual); Study Completion 2025-12-28 (Actual)

PRIMARY OUTCOMES:
Cancer Fatigue Scale | 30 days
  A five-point Likert scale (1-5) is used for each question. Cronbach's alpha value was 0.74. The scale consists of "physical" (7 items) (1,2,3,6,9,12,15), "cognitive" (4 items) (4,7,10,13), "emotional" (4 items) (5,8,11,14), 3 subheadings and 15 questions in total. In the analysis of the scale, physical state (item 1+2+3+6+9+12+15) is calculated by subtracting 7 from the total, emotional state (item 5+8+11+14) is calculated by adding, cognitive state (item 4+7+10+13) is calculated by subtracting 4 from the total. The total score is calculated by summing the physical, emotional and cognitive states. The minimum score is 4 and the maximum score is 64.
Chemotherapy-Induced Peripheral Neuropathy Assessment Tool | 30 days
  The first 6 questions in the scale are sensory symptoms and questions 7-9 are motor symptoms sub-dimensions. Experiencing the symptom of peripheral neuropathy (1=Yes, 2=No), the severity of the symptom (1=Never severe, 10= Extremely severe), the distress caused by the symptom (1= Never caused, 10= Extremely caused), the frequency of the symptom (1= Never experienced, 10= Continuously experienced), the activities of peripheral neuropathy symptoms (1= Never prevented, 10= Completely prevented). The first 9 items assess symptom presence (0-1), symptom severity (0-10), emotional distress (0-10) and frequency (0-10). The total score that can be obtained from the scale is between 0-279.
Trait Anxiety Inventory | 30 days
  The reversed statements of the Trait Anxiety Inventory (SAI) consist of items 21, 26, 27, 30, 33, 36 and 39. A total score between 20 and 80 is obtained from the scale. After the total scores of the direct and inverted statements are found separately, the total score obtained for the direct statements is subtracted from the total score obtained for the inverted statements. A predetermined and unchanging value is added to this number. This value is 35 for the SDI. The last value obtained is the anxiety score of the individual. A low score means that the anxiety level of the individual is low and a high score means that the anxiety level of the individual is high.

CONTACTS AND LOCATIONS:
Overall Officials: Naciye Esra koyuncu, Study Chair — NECMETTİN ERBAKAN ÜNİVERSİTESİ SB ENSTİTÜSÜ
Locations (1):
- Necmettin Erbakan University, Konya, Meram, Turkey (Türkiye)

REFERENCES:
- [Result] Alejandro LM, Behrendt CE, Chen K, Openshaw H, Shibata S. Predicting acute and persistent neuropathy associated with oxaliplatin. Am J Clin Oncol. 2013 Aug;36(4):331-7. doi: 10.1097/COC.0b013e318246b50d. PMID 22547012